CLINICAL TRIAL: NCT06377618
Title: Comparison Of Resistance Training And Core Strengthening Exercises Along With Vitamin D Intake In Postmenopausal Women With Low Back Pain
Brief Title: Comparison Of Resistance Training And Core Strengthening Exercises Vitamin D In Postmenopausal Women With Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/556
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Menopausal; Pain, Low Back
MeSH Terms: conditions — Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training and Core Strengthening Exercises Group (Experimental): The regimen includes resistance training (using bands, weights, and bodyweight for major muscle groups) and core strengthening (targeting abdominal, lower back, hip, and gluteal muscles) exercises.
  Interventions: Diagnostic Test: Resistance Training and Core Strengthening Exercises Group
- Resistance Training and Core Strengthening Exercises Group Plus Vitamin D Supplementation (Other): Identical exercise protocol to Group 1, with three supervised sessions per week.
  First Arm Intervention plus Vitamin D Supplementation: Daily vitamin D supplementation, with the dosage adjusted based on initial serum 25(OH)D levels to achieve and maintain optimal vitamin D status. Typical dosages range from 800 to 2000 IU/day, subject to adjustments as necessary.
  Serum 25(OH)D levels and potential supplementation-related adverse effects will be monitored at baseline and after 12 weeks.
  Outcome Measures: In addition to the same outcome measures as Group 1, changes in serum 25(OH)D levels will also be assessed.
  Interventions: Diagnostic Test: Resistance Training and Core Strengthening Exercises Group Plus Vitamin D Supplementation

INTERVENTIONS:
Diagnostic Test: Resistance Training and Core Strengthening Exercises Group — The regimen includes resistance training (using bands, weights, and bodyweight for major muscle groups) and core strengthening (targeting abdominal, lower back, hip, and gluteal muscles) exercises.
  Arms: Resistance Training and Core Strengthening Exercises Group
Diagnostic Test: Resistance Training and Core Strengthening Exercises Group Plus Vitamin D Supplementation — Group 1 Intervention plus Vitamin D Supplementation: Daily vitamin D supplementation, with the dosage adjusted based on initial serum 25(OH)D levels to achieve and maintain optimal vitamin D
  Arms: Resistance Training and Core Strengthening Exercises Group Plus Vitamin D Supplementation

SUMMARY:
This study aims to evaluate the effectiveness of resistance training, core strengthening exercises, and vitamin D supplementation in reducing low back pain (LBP) among postmenopausal women.

DETAILED DESCRIPTION:
Postmenopausal women are particularly susceptible to LBP due to physiological changes such as reduced estrogen levels, decreased muscle mass, and bone density. The randomized controlled trial (RCT) will be conducted over six months in various clinical settings in Lahore, with a sample size of 36 participants, divided into two groups. The inclusion criteria focus on postmenopausal women aged 50-70 years experiencing LBP for at least three months and who are not currently taking vitamin D supplements. Data on pain intensity, functional disability, muscle strength, endurance, and vitamin D levels will be collected and analyzed to assess the interventions' impact. The study's findings could provide evidence-based recommendations for managing LBP in postmenopausal women, combining physical activity with nutritional supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50-70 years.
* Experiencing low back pain for at least 3 months.
* Capable of engaging in light to moderate physical exercise.

Exclusion Criteria:

* History of spinal surgery.
* currently taking vitamin D supplements.
* Diagnosed with severe osteoporosis.
* Chronic use of pain medication that cannot be temporarily ceased.
* Current participation in another clinical trial.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6 Month
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable
Oswestry Disability Index (ODI) | 6 Months
  a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan